CLINICAL TRIAL: NCT03261388
Title: ABLE POWER - Activity Based Locomotor Exercise PrOgram: Wait-list controllEd Research
Brief Title: Activity Based Locomotor Exercise PrOgram-Wait-list controllEd Research
Acronym: ABLE-POWER
Status: Terminated | Type: Observational
Why Stopped: Change in subject population/ABLE POWER program
Sponsor: Allina Health System (Other)
Responsible Party: Principal Investigator, Nancy Flinn, Senior Scientific Advisor, Allina Health System
Other Study IDs: CK-1604
Record Dates: First submitted 2017-08-17; First posted 2017-08-25 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ABLE POWER Program: Participants on the Activity-Based Locomotor Exercise Program (ABLE) waitlist will be enrolled prior to beginning the ABLE program. This waiting period will allow outcomes to be compared (in the same participant) before receiving the intervention and after receiving the intervention.
  Interventions: Behavioral: Activity-Based Locomotor Exercise Program (ABLE)

INTERVENTIONS:
Behavioral: Activity-Based Locomotor Exercise Program (ABLE) — The ABLE program is an intensive locomotor based intervention that is offered at the Golden Valley Courage Kenny Rehabilitation Institute.

SUMMARY:
At Courage Kenny Rehabilitation Institute, rehabilitation for individuals with spinal cord injury (SCI) is being led by the NIH funded NeuroRecovery Network (NRN) Community Fitness and Wellness Program through the Activity-Based Locomotor Exercise Program (ABLE). Any individual with a spinal cord injury who is eligible for the ABLE Program is eligible for participation in the NeuroRecovery Network Research Project (NRN). The purpose of the ABLE POWER Study is to evaluate the effectiveness of activity-based locomotor exercise programs in individuals with SCI through a wait-list controlled design. Individuals who have a spinal cord injury and are on the wait list for ABLE will be enrolled in this project for a year while they wait for an opening in the ABLE program. Changes that occur while participants are on the wait list will be compared to changes that occur after they are enrolled in ABLE. A difference in the rate of improvement after enrollment in the intervention would be attributed to the ABLE intervention. Individuals participating in the ABLE program will receive the ABLE intervention regardless of participation in the ABLE POWER research study. In this design, there will be two measures in the year prior to enrollment in ABLE, and two measures in the year after enrollment, and the two time periods would be compared to the data collected at enrollment into ABLE.

ELIGIBILITY:
Inclusion Criteria:

* The participant must be eligible for the Neurorecovery Network (NRN) Study. Eligibility criteria for the NRN study are as follows: The participant must have a spinal cord injury, at any spinal level or time since injury. Individuals with uncontrolled diabetes, uncontrolled seizures, uncontrolled autonomic dysreflexia, uncontrolled hypotension, unstable angina, history of heart attack, osteoporosis, or weight of more than 275 pounds (due to the weight limit of the partial weight supported treadmill system) are not eligible.
* The participant must be on the ABLE wait list.

Exclusion Criteria:

• The participant must NOT have previously participated in ABLE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for this research study will be recruited from adults with spinal cord injury (SCI) on the wait list for the Neurorecovery Network (NRN) research study. These individuals have injuries at all spinal levels and categories of completeness.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Change in Neuromuscular Recovery Scale (NRS) | At entry to wait list, after 6 months, at enrollment to the ABLE program (6-13 months after entry to wait list), 6 months post entry to ABLE, 12 months post entry to ABLE
  The NRS measures motor function in individuals with SCI without allowing compensatory motions. This 15 item measure is collected while the participants are on the mat, in sitting, standing, and on the weight supported treadmill. Items include upper extremity function, lower extremity function, sitting, sit to stand, standing, and locomotor items.

SECONDARY OUTCOMES:
Change in Canadian Occupational Performance Measure (COPM) | At entry to wait list, after 6 months, at enrollment to the ABLE program (6-13 months after entry to wait list), 6 months post entry to ABLE, 12 months post entry to ABLE
  The COPM is a client-centered measure of performance and satisfaction using client identified meaningful activities and has been used with individuals who have SCI as a means to identify personally meaningful goals
Change in Craig Handicap Assessment and Reporting Technique (CHART) | At entry to wait list, after 6 months, at enrollment to the ABLE program (6-13 months after entry to wait list), 6 months post entry to ABLE, 12 months post entry to ABLE
  The Craig Handicap Assessment and Reporting Technique (CHART) is a measure of social participation in individuals with SCI.
Change in American Spinal Injury Association Impairment Scale (AIS) | At entry to wait list, at enrollment to the ABLE program (6-13 months after entry to wait list), 12 months post entry to ABLE
  The American Spinal Injury Association Impairment Scale (AIS) classifies the motor and sensory impairment that results from a SCI, and is the gold standard for identifying completeness of a SCI.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Flinn, PhD, OTR/L, Principal Investigator — Allina Health
Locations (1):
- Courage Kenny Rehabilitation Institute, Golden Valley, Minnesota, United States